CLINICAL TRIAL: NCT00146224
Title: A Randomized, Double-Blind, Equivalence Study of the Efficacy of Epoetin Alfa Manufactured by Deep Tank Bioreactor Technology and Epoetin Alfa Manufactured by Roller-Bottle Technology for the Treatment of Anemia in Patients With Chronic Kidney Disease (CKD) Receiving Hemodialysis
Brief Title: Efficacy of Epoetin Alfa Deep Tank in Treatment of Anemia in Patients With Chronic Kidney Disease Receiving Hemodialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20050113
Record Dates: First submitted 2005-09-06; First posted 2005-09-07 (Estimated); Last update posted 2010-02-26 (Estimated); Status verified 2010-02

CONDITIONS: Nephrology
Keywords: anemia; chronic kidney disease, CKD; hemodialysis; epoetin; Epogen®
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — Epoetin Alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Epoetin alfa RB (Active Comparator)
  Interventions: Drug: Epoetin alfa RB
- Epoetin alfa DT (Experimental)
  Interventions: Drug: Epoetin alfa DT

INTERVENTIONS:
Drug: Epoetin alfa RB — Receive drug at same frequency and dose as at the time of randomization Change dose by+/- 25% in order to maintain Hb between 10.0 - 13.0 g/dL and within -1.0 to +1.5 g/dL of the subject's baseline Hb.
  Arms: Epoetin alfa RB
Drug: Epoetin alfa DT — Receive drug at same frequency and dose as at the time of randomization Change dose by+/- 25% in order to maintain Hb between 10.0 - 13.0 g/dL and within -1.0 to +1.5 g/dL of the subject's baseline Hb.
  Arms: Epoetin alfa DT

SUMMARY:
The purpose of this study is to evaluate whether the efficacy of Epoetin alfa DT is equivalent to that of Epoetin alfa RB for the treatment of anemia in patients with CKD receiving hemodialysis

ELIGIBILITY:
Inclusion Criteria: - Diagnosis of CKD and receiving hemodialysis for greater than or equal to 3 months before randomization - Mean HB level between 10 and 13 g/dL (inclusive) (mean of 2 values drawn at least 3 days apart during the screening period) - Currently receiving a stable dose of Epoetin alfa RB (i.e., EPOGEN® or PROCRIT®) for at least 6 weeks prior to randomization. Stable is defined as: less than or equal to 25% change in dose over 6 weeks, same frequency and route of administration with no more than 1 missed or withheld dose during each of the two three-week periods before randomization Exclusion Criteria: - Uncontrolled hypertension, defined as a pre-dialysis systolic BP greater than 180 and/or diastolic BP of greater than 110 during the screening period - Known history of severe hyperparathyroidism (PTH Greater than 1500 pg/ml within 3 months prior to enrollment) - Currently receiving immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2005-09; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Ratio of weekly dose at the evaluation period to the weekly dose at baseline | Entire Study
Change in Heloglobin level between the screening period and the evaluation period | Entire Study

SECONDARY OUTCOMES:
Change from baseline Hb at each measurement timepoint | Entire Study
Maintaining Hemoglobin within range at each measurement timepoint | Entire Study
Average Epoetin alfa dose over evaluation period | evaluation period (weeks 21 - 28)
Change from baseline dose at each measurement timepoint | entire study
Epoetin alfa seroreactivity | entire study
Subject incidence, nature and severity of adverse events | entire study
Hemoglobin variability | entire study
changes from baseline laboraotry and vital sign parameters | entire study

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Lei L, Olson K. Evaluating statistical methods to establish clinical similarity of two biologics. J Biopharm Stat. 2010 Jan;20(1):62-74. doi: 10.1080/10543400903115082. PMID 20077249
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_05_EPO_20050113.pdf
- See also: FDA-approved Drug Labeling — http://www.epogen.com/